CLINICAL TRIAL: NCT06724471
Title: Preservation of Women's Fertility: Evaluation of Innovative Methods for Ovarian Tissue Cryopreservation
Acronym: FERTIOVO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: CryoBioSystem (Unknown); IMoST UMR 1240 Inserm-Université Clermont Auvergne (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022_Brugnon_FERTIOVO
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Infertility, Female
Keywords: Human ovarian tissue; Cryopreservation; Fertility Preservation; Organotypic culture; Female infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Fresh ovarian cortex fragments: Pericystic ovarian cortex will be cut into 1mm3 fragments and either directly analyzed on the day of collection (D0) or after organotypic culture (D7 and D14).
- Fragments of ovarian cortex frozen in thermosoldered cryovials.: Pericystic ovarian cortex will be cut into 1mm3 fragments, frozen using a slow programmable freezing device (Nano Digitcool, Cryo Bio System) in thermosoldered cryovials and stored in liquid nitrogen (-196°C). Then, fragments will be thawed before being analyzed on the day of thawing (D'0) and after 7 and 14 days (D7 and D14) of organotypic culture.
  Interventions: Device: Human ovarian tissue cryopreservation using thermosoldered or screwed cryovials
- Fragments of ovarian cortex frozen in screwed cryovials.: Pericystic ovarian cortex will be cut into 1mm3 fragments, frozen using a slow programmable freezing device (Nano Digitcool, Cryo Bio System) in screwed cryovials and stored in liquid nitrogen (-196°C). Then fragments will be thawed before being analyzed on the day of thawing (D'0) and after 7 and 14 days (D7 and D14) of organotypic culture.
  Interventions: Device: Human ovarian tissue cryopreservation using thermosoldered or screwed cryovials

INTERVENTIONS:
Device: Human ovarian tissue cryopreservation using thermosoldered or screwed cryovials — Human ovarian tissue Cryopreservation: immediately after cyst resection, pericystic ovarian cortex will be cut into 1mm3 fragments and cryopreserved in screwed or thermosoldered cryovials using a slow programmable freezing device (Nano Digitcool, Cryo Bio System).
  Groups: Fragments of ovarian cortex frozen in screwed cryovials.; Fragments of ovarian cortex frozen in thermosoldered cryovials.

SUMMARY:
The recent innovations in cancer diagnosis and therapy have improved the five-year survival for patients. However, anticancer treatments may impair patient fertility; therefore fertility preservation is recommended before therapy initiation. The sole method for preserving young prepubescent girls' fertility, which can also be used for pubescent women, is ovarian tissue cryopreservation (OTC) with later auto-transplantation. Although 200 births have been reported worldwide after OTC and transplantation, significant improvements are required. Indeed, freezing and thawing protocols vary according to laboratories (media, cryoprotectants, freezing curve, etc…) and selection criteria are not justified. In addition, most of the laboratories use unsafe devices (e.g. screw cap cryovials) for OTC, exposing ovarian tissues to biological hazards during sample storage in nitrogen tanks. To eliminate these risks, novel "high security" devices have been commercialized (welded cryotubes). However, while thermal welding could alter tissue quality, the functionality of the human ovarian tissue frozen with these innovative devices has not yet been evaluated. The objectives of this study are i) to optimize the freezing and the thawing protocols for human OTC according to thermodynamic properties of the freezing medium and the type of device (welded or screwed cryotube) and ii) to determine if the type of cryotube influences the quality of human ovarian tissue.

This project will enable to reach a better understanding of the impact of freezing on ovarian tissue functionality, as well as the implementation of an optimal protocol for OTC within the ART laboratory of Clermont-Ferrand hospital to optimize patient care.

DETAILED DESCRIPTION:
The aim of this project is to determine whether the type of cryogenic tube (with screw caps or thermosoldered) influences the quality and functionality of ovarian tissue after cryopreservation. First, a characterization of the thermodynamic properties of the freezing medium using a differential scanning calorimeter (Diamond DSC, PerkinElmer) will be carried out to optimize freezing and thawing protocols. This analysis will define important parameters such as crystallization temperature (Tc), end-of-melting temperature (Tm), and transition temperatures (Tg'1). Once freezing and thawing protocols are optimized, the investigators will use human ovarian cortex surrounding benign cysts, a model previously validated by our laboratory, to determine whether the type of cryotube influences the quality of human ovarian tissue. These ovarian cortical samples usually destroyed in clinics share similar characteristics with normal ovarian cortex. Ovarian tissue will be cut into 1mm3 fragments and divided into three groups: fresh ovarian cortex (group1, control), ovarian cortex cryopreserved in thermosoldered cryogenic tubes (group 2) or in screw cap (group 3). The investigators will assess ovarian tissue quality immediately after resection for group 1 or after thawing for group 2 and 3 by analyzing follicle density and morphology (HES staining) and proliferation/apoptosis balance (Immunohistochemistry (IHC) for KI67 and cleaved caspase 3). To assess the functionality of the ovarian tissue after thawing, ovarian cortex fragments will be in vitro cultured. The investigators will analyze i) follicle density, type and morphology (HES staining), ii) the proliferation/apoptosis balance (IHC for KI67 and cleaved caspase 3), iii) the expression levels of major folliculogenesis regulators (IHC for GDF-9) and iv) the levels of folliculogenesis-associated hormones (AMH, estrogen) secreted in culture medium.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman scheduled for benign ovarian cyst resection (dermoid, functional, mucinous or serous cysts)
* Below 37 years old and above 18 years old
* Capable of giving written informed consent to participate in the research study
* Affiliated to social welfare service

Exclusion Criteria:

* Women above 37 years old and below 18 years old
* Polycystic ovary syndrome
* Diminished ovarian reserve
* Severe endometriosis
* Malignant and endometrial cysts

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult woman scheduled for benign ovarian cyst resection in the University Hospital Center of Clermont-Ferrand.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-thawing Ovarian Follicle morphology | 24 months
  Follicle morphology of fresh versus frozen (with thermosoldered or screwed cryovials)/thawed ovarian cortex will be assessed on serial sections stained with hematoxylin-eosin-saffron. Fragments will be fixed on the day of collection for group 1 and directly after thawing for groups 2 and 3. Morphology of follicles will be evaluated according to the parameters described by Keros et al. Hum Reprod. 2009.

SECONDARY OUTCOMES:
Post-thawing Ovarian Follicle density | 24 months
  Follicle density (=number of follicle/mm2) of fresh versus frozen (with thermosoldered or screwed cryovials)/thawed ovarian cortex will be assessed on serial sections stained with hematoxylin-eosin-saffron. Fragments will be fixed on the day of collection for group 1 and directly after thawing for groups 2 and 3.
Post-thawing Ovarian Follicle proliferation | 24 months
  the percentage of proliferative (oocyte or granulosa cells positive for KI-67 in fresh and frozen (with thermosoldered or screwed cryovials) /thawed ovarian cortex will be assessed on immunostained serial sections. Fragments will be fixed on the day of collection for group 1 and directly after thawing for groups 2 and 3.
Post-thawing Ovarian Follicle apoptosis | 24 months
  the percentage of apoptotic (oocyte or granulosa cells positive cleaved caspase 3) in fresh and frozen (with thermosoldered or screwed cryovials) /thawed ovarian cortex will be assessed on immunostained serial sections. Fragments will be fixed on the day of collection for group 1 and directly after thawing for groups 2 and 3.
Ovarian Follicle stage after organotypic culture | 36 months
  Follicle stages (% of primordial, primary, secondary and antral follicles) in fresh versus frozen (with thermosoldered or screwed cryovials)/thawed ovarian cortex will be assessed on serial sections stained with hematoxylin-eosin-saffron. Fragments will be fixed after 7 or 14 days of organotypic culture.
Ovarian Follicle morphology after organotypic culture | 36 months
  Follicle morphology of fresh versus frozen (with thermosoldered or screwed cryovials)/thawed ovarian cortex will be assessed on serial sections stained with hematoxylin-eosin-saffron. Fragments will be fixed after 7 or 14 days of organotypic culture. Morphology of follicles will be evaluated according to the parameters described by Keros et al. Hum Reprod. 2009.
GDF-9 expression after organotypic culture | 36 months
  the percentage of GDF9 positive follicles (i.e. with an oocyte positive for GDF-9) in fresh and frozen (with thermosoldered or screwed cryovials) /thawed ovarian cortex will be assessed on immunostained serial sections. Fragments will be fixed after 7 or 14 days of organotypic culture.
Proliferation after organotypic culture | 36 months
  the percentage of proliferative (oocyte or granulosa cells positive for KI-67) in fresh and frozen (with thermosoldered or screwed cryovials) /thawed ovarian cortex will be assessed on immunostained serial sections. Fragments will be fixed after 7 or 14 days of organotypic culture.
Apoptosis after organotypic culture | 36 months
  the percentage of apoptotic (oocyte or granulosa cells positive cleaved caspase 3) in fresh and frozen (with thermosoldered or screwed cryovials) /thawed ovarian cortex will be assessed on immunostained serial sections. Fragments will be fixed after 7 or 14 days of organotypic culture.
AMH secretion after organotypic culture | 36 months
  AMH levels will be quantified in culture medium during organotypic culture of fresh and frozen (with thermosoldered or screwed cryovials) /thawed ovarian cortex. Culture media will be harvested every three days of culture for 14 days. AMH will be quantified by electrochemiluminescence
Estrogen secretion after organotypic culture | 36 months
  Estrogen levels will be quantified in culture medium during organotypic culture of fresh and frozen (with thermosoldered or screwed cryovials) /thawed ovarian cortex. Culture media will be harvested every three days of culture for 14 days. Estrogen will be quantified by electrochemiluminescence
Thermodynamic properties of freezing medium | 12 months
  A differential scanning calorimeter (DiamondDSC, PerkinElmer) will be used to determine the crystallization temperature (Tc), end-of-melting temperature (Tm), and transition temperature (Tg'1) of the freezing medium (Leibovitz with 4 mg/mL HSA, 1.5M DMSO and 0.1M sucrose).

CONTACTS AND LOCATIONS:
Overall Officials: Florence Brugnon, MD, PhD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- University Hospital, Clermont-Ferrand, France